CLINICAL TRIAL: NCT05893836
Title: Real-World Disease Management and Outcomes in Chronic Myeloid Leukaemia
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001AGB01
Record Dates: First submitted 2023-05-17; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Chronic myeloid leukaemia (CML) diagnosis is based on the demonstration of a BCR-ABL fusion transcript expressed by the Philadelphia (Ph) chromosome by RQ-PCR and/or the demonstration of t(9;22)(q34;q11) by conventional karyotyping or interphase FISH. As per standard practice, response to therapy is monitored using either molecular or cytogenetic tests or both; specifically, patients are monitored by quantitative PCR on peripheral blood, supplemented by bone marrow karyotyping if it was clinically indicated. ABL kinase mutational analysis is carried out when the transcript ratio has increased over two sequential samples or on clinical demand. Testing for T315I mutation is also performed for patients who fail to respond to first line TKI and all patients who acquire TKI resistance over the course of their treatment.

Data collection is initiated six months after date of diagnosis; research nurses working to agreed operating procedures and data standards visit each of the 14 hospitals in the region and abstract a core clinical dataset from the patients' medical records. The information collected includes demographic details, baseline blood count data and first line treatment. All details are abstracted onto structured forms and entered onto the web-based system, which integrates Haematological Malignancy Research Network (HMRN) and Haematological Malignancy Diagnostic Service (HMDS) data. An important feature of data acquisition is the emphasis on primary source information; data from radiology reports, blood tests, clinical examination, and clinician summaries are recorded, enabling embedded algorithms in the database system to automatically generate stage and prognostic scores. Further data abstraction from the medical records has been undertaken to capture information on subsequent treatment lines. Information on date and cause of death were obtained from the National Health Service (NHS) Central Register.

ELIGIBILITY:
Inclusion Criteria:

• Adult (18+ years) patients newly diagnosed with CML in chronic phase (ICD-O-3: 9875/3) by HMDS between 1st September, 2004 to 31st August, 2019 whilst resident in the HMRN region and treated within the Network.

Exclusion Criteria:

None specified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who received tyrosine kinase inhibitors (TKIs), by treatment llne | Up to 18 years
Year treatment started, by TKI | Up to 18 years

SECONDARY OUTCOMES:
Number of patients with response to TKIs | Up to 12 months
  Disease response was defined as either a major molecular response (MMR, ≤ 0.1% BCR-ABL1) or as an MR2, which is a molecular response (MR, ≤ 1.0% BCR-ABL1), or complete cytogenetic remission (CCyR).
Time to response to TKIs | Up to 12 months
Reason for switching TKI | Up to 12 months
Number of patients tested for T315I mutation by treatment line | Up to 12 months
Overall survival (OS) | Up to 10 years
  OS was defined as the time (in years) from initiation of treatment (i.e., the index date) to death (any cause).
Progression-free survival | Up to 10 years
  PFS was defined from the initiation of treatment (i.e., the index date) to the earliest documentation of disease progression to accelerated phase/blast crisis (AP/BC) or date of death from any cause.
Time to treatment discontinuation | Up to 10 years
Relative survival by treatment line | Up to 10 years
  Relative survival (RS) was estimated to examine the CML-specific mortality rate. The Stata program strel (v1.2.7) was used to estimate RS and corresponding 95% Confidence Intervals (95%CI); with age and sex-specific background mortality rates being obtained from national life tables.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Haematological Malignancy Research Network, York, United Kingdom